CLINICAL TRIAL: NCT06202911
Title: Effect of Oral N-Acetyl Cysteine in Prevention of Necrotizing Enterocolitis in Preterm Neonates With Feeding Intolerance
Acronym: Oral NAC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ekram Hassan
Record Dates: First submitted 2023-12-23; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-12

CONDITIONS: Preterm Neonates and Feeding Intolerance; Necrotizing Enterocolitis; Oral N-acetyl Cysteine
Keywords: preterm neonates; neonates; feeding intolerance; necrotizing enterocolitis; prematurity; n-acetyl cysteine; oral n-acetyl cysteine
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- intervention group (Active Comparator): preterm neonates with feeding intolerance, pre-Nec., receive the drug
  Interventions: Drug: oral n-acetyl cysteine
- control group (Placebo Comparator): preterm neonates
  Interventions: Other: placebo

INTERVENTIONS:
Drug: oral n-acetyl cysteine — the active participants will receive oral N-acetyl cysteine with dose 20mg/dose every 6 hours for 10 days or until reaching full feeding or resolution of feeding intolerance
  Arms: intervention group
Other: placebo — the control group will receive placebo
  Arms: control group

SUMMARY:
necrotizing enterocolitis is a dangerous disease that may be fatal especially in preterm neonates, the early features of the disease are symptoms of feeding intolerance and interruption of the baby's feeding plan , so prophylactic measures at this stage may help to prevent its progression and its complications.

N-acetyl cysteine is an FDA- approved drug and has many uses in different diseases and in different age groups including neonates, it has a mucolytic and anti-inflammatory and anti-oxidant effects that are believed to break the bacterial biofilm which enables it to stick to the intestinal wall and also decrease the intestinal wall inflammation, therefore enhance the intestinal barrier and decrease the chance of bacterial invasion.

ELIGIBILITY:
Inclusion Criteria:

* preterm neonates (less than or = 36 weeks gestational age )
* feeding intolerance

Exclusion Criteria:

* active gastro-intestinal tract bleeding
* Gastro- intestinal tract surgical problem
* Congenital gastro-intestinal tract anomalies
* evidence of allergy to NAC
* use of prebiotics or probiotics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
incidence of necrotizing enterocolitis | 10 days
  assess the development of necrotizing enterocolitis

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
for patient confidentiality

REFERENCES:
- [Background] undefined
- See also: Related Info — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&q=N-acetyl+cysteine+may+prevent+severe+intestinal+damage+in+necrotizing+enterocolitis&btnG=